CLINICAL TRIAL: NCT01613495
Title: Ghrelin Suppression by Sandostatin LAR® Depot (Octreotide Acetate for Injectable Suspension) in Patients With Prader-Willi Syndrome
Brief Title: Ghrelin Suppression by Octreotide in Prader-Willi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan Purnell, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: eIRB #1265; OCTRI # __910_____ (Other: Oregon Health and Sciences University)
Record Dates: First submitted 2011-04-13; First posted 2012-06-07 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Prader Willis Syndrome
Keywords: obesity
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity | interventions — Saline Solution; Octreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo
- Octreotide (Active Comparator): They will be admitted to the inpatient unit of the OCTRI for testing six times. During each of these visits, testing will include measuring how well glucose (sugar) is processed, how much energy is burned off as heat, their amount of body fat, levels of the hormone ghrelin, and how much food is eaten at a meal. After the first study visit, subjects will begin monthly treatment with either the study drug or a placebo (an inactive substance), which will be continued for the first six months of the study. For the last six months of the study, subjects will be switched to the opposite treatment. During these study periods participants will return monthly for administration of study medication, physical examination, and blood draw to check liver enzymes.
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Placebo — After the first study visit, subjects will begin monthly treatment with either the study drug or a placebo (an inactive substance), which will be continued for the first six months of the study. For the last six months of the study, subjects will be switched to the opposite treatment. During these study periods participants will return monthly for administration of study medication, physical examination, and blood draw to check liver enzymes.
  Other Names: Normal Saline
  Arms: Placebo
Drug: Octreotide — They will be admitted to the inpatient unit of the OCTRI for testing six times. During each of these visits, testing will include measuring how well glucose (sugar) is processed, how much energy is burned off as heat, their amount of body fat, levels of the hormone ghrelin, and how much food is eaten at a meal. After the first study visit, subjects will begin monthly treatment with either the study drug or a placebo (an inactive substance), which will be continued for the first six months of the study. For the last six months of the study, subjects will be switched to the opposite treatment. During these study periods participants will return monthly for administration of study medication, physical examination, and blood draw to check liver enzymes.
  Other Names: Sandostatin
  Arms: Octreotide

SUMMARY:
The purpose of this study is to learn more about how octreotide (Sandostatin LAR® Depot) affects levels of ghrelin, hunger, and body weight in people with Prader-Willi Syndrome.

DETAILED DESCRIPTION:
After baseline tests, a nurse will administer monthly injections of Sandostatin LAR® or placebo for 6 months. At the end of this initial 6-month treatment period and a 4-month washout period, study subjects will then crossover to receive the alternative therapy (placebo or octreotide) for an additional 6 months. Subjects will be followed for 16 months total at scheduled visits: 0, 2, 6, 10, 12, and 16 months (Table 2).

ELIGIBILITY:
Inclusion Criteria:

* o Diagnosis of PWS confirmed by chromosome analysis (i.e. interstitial deletion of paternally-derived chromosome 15Q, uniparental maternal disomy or other chromosome 15 abnormalities)

  * Age 18 years and older
  * Written informed consent obtained (by subject or guardian) and willingness to comply with the study schedule and procedures
  * Free T4, TSH values in the normal range (with or without thyroxine replacement)
  * Subjects with confirmed hypogonadism who are corrected with adequate doses of sex steroid replacement, will have been treated for at least 6 months prior to entry and have no change in dosages over the study period.
  * Patients with confirmed growth hormone deficiency who are corrected with adequate doses of replacement, will have been treated for at least 6 months prior to entry and have no change in dosages over the study period.

Exclusion Criteria:

* Symptomatic gallstones.
* Smokers.
* Alcohol consumption > 2 drinks per day.
* Exercise > 30 minutes 3 times a week.
* Weight > 500 lbs (exceeds the limit for the BODPOD).
* Active pulmonary infection.
* Sleep disorder.
* Subjects will be excluded if they have clinically significant disease that would have an impact on metabolic outcomes or body composition including diabetes mellitus, chronic inflammatory bowel disease, chronic severe liver or kidney disease, heart disease, cancer, symptomatic gallstones, or neurological disorders
* history of hepatic disease (patients with minimal, i.e., <3Xs the upper limit of normal for LFTs indicative of hepatic steatosis, MAY participate)
* pregnant or lactating
* known hypersensitivity to Sandostatin acetate or other related drug or compound
* subjects who exhibit symptoms indicative of intolerance following the 100 mcg test dose of Sandostatin Injection, SC
* subjects who have previously received Sandostatin® (octreotide)
* subjects who have received other investigational drugs administered or received within 30 days of study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-08; Primary Completion 2024-03 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Ghrelin levels | Change from baseline to 6 months
Appetite | Change from baseline to 6 months
Body weight | Change from baseline to 6 months

SECONDARY OUTCOMES:
Hormone levels | Change from baseline to 6 months
Body composition | Change from baseline to 6 months
Energy expenditure | Change from baseline to 6 months
Glucose metabolism | Change from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q Purnell, M.D., Principal Investigator — Oregon Health and Science University; Jonathan Q Purnell, M.D., Principal Investigator — Oregon Health & Sciences University Portland, OR